CLINICAL TRIAL: NCT04775888
Title: Prophylaxis and On-demand Treatment for Persons With Haemophilia and Other Coagulation Deficiencies: a Comparison of Perceived and Observed Accessibility in the Auvergne-Rhône-Alpes Region (France)
Brief Title: Accessibility of Prophylaxis and On-demand Treatment for Persons With Haemophilia and Other Coagulation Deficiencies
Acronym: PHAREO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RESCUe - RESeau Cardiologie Urgence / RESUVal - RESeau des Urgences de la vallée du Rhône (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PHAREO
Record Dates: First submitted 2021-02-11; First posted 2021-03-01 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-02

CONDITIONS: Health Services Accessibility; Blood Coagulation Factor Deficiencies
Keywords: haemophilia; accessibility; on-demand treatment; prophylactic treatment
MeSH Terms: conditions — Coagulation Protein Disorders; Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current treatment of people with haemophilia and other bleeding deficiencies is largely based on clotting factor replacement therapy. The injections can be repeated several times a week according to a personalized schedule. To date, medications are exclusively dispensed in hospital pharmacies to ensure traceability and safety. This retrocession imposes accessibility constraints on patients and on their caregivers, increasing the burden of the disease, particularly in the organization of personal and professional daily life. The PHAREO study aims to investigate patients' perception of accessibility to anti-haemophilia drugs in relation to an evaluation of spatial accessibility in the Auvergne-Rhône-Alpes region (France) in order to consider, if necessary, ways of improving the pathway for patients and their caregivers.

DETAILED DESCRIPTION:
Haemophilia is a rare constitutional hemorrhagic disease whose drug management is based on the use of chronic lifelong replacement therapy. For many years, the reference treatment, particularly in children, has been based on the use of anti-haemophilic drugs for prophylaxis requiring repeated injections several times a week according to a personalized schedule. In contrast, on-demand treatment is less and less used, particularly in patients with severe forms of haemophilia. Clinical and biological diagnosis, as well as the implementation and monitoring of treatments, are carried out within specialized hospital care structures affiliated with the French national reference center. Medications are dispensed as part of hospital retrocessions. This organization imposes constraints on patients and their caregivers due to their limited accessibility.

The burden related to this disease is probably due to the systematic use of specialized hospital teams such as doctors, nurses for self-injection training for example, and pharmacists. It now seems important to reflect on the evolution of patient pathways that were previously exclusively hospital-centred towards ambulatory care. To do this, various reflections need to be undertaken, including that relating to the accessibility of medication. Indeed, the monthly renewals of these chronic treatments force patients and their caregivers, as well as the parents of children, to go to the hospital, which frequently makes the organization of daily and professional life more cumbersome.

The PHAREO study aims to investigate patients' perception of accessibility to anti-haemophilia drugs in relation to an evaluation of spatial accessibility in order to consider, if necessary, ways of improving the pathway for patients and their caregivers.

The expected benefits of the study are to have: 1) an exhaustive description of the spatial accessibility of the cohort of people living with haemophilia to anti-haemophilia medication within the Auvergne Rhône Alpes region (France) and 2) a better understanding of their needs and their perceptions regarding access to on-demand and prophylactic treatments.

ELIGIBILITY:
Included:

* Living person on the study start date and presenting with haemophilia or other coagulation deficiencies;
* Treated with prophylaxis or on-demand anti-haemorrhagic treatments;
* Location of medication dispensing within the hospital pharmacies of the HEsora network (Hémophilie Soins Rhône Alpes): 27 eligible hospital pharmacies in Rhône Alpes + <10 eligible hospital pharmacies in Auvergne

Excluded:

- Home delivery (not included in the study via hospital pharmacy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The included subjects comprise people with haemophilia or other coagulation deficiencies, with no limitation of age, treated by prophylaxis or on-demand treatment, in one of the authorized hospital pharmacies in the Auvergne-Rhone-Alpes region (France).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-21 (Estimated)

PRIMARY OUTCOMES:
To assess the perception of persons with haemophilia and other coagulation deficiencies regarding the accessibility to prophylactic and on-demand antihemorrhagic treatment | Through study completion, on average 6 months.
  The perception is defined by the satisfaction level of the survey participants, measured with on item in the questionnaire (Very satisfied / Rather satisfied / Rather not satisfied / Not satisfied).
To measure the accessibility of persons with haemophilia and other coagulation deficiencies regarding the accessibility to prophylactic and on-demand antihemorrhagic treatment | Through study completion, on average 6 months.
  The accessibility is measured by spatial analysis, representing the distance between the home and/or work zip codes and the hospital pharmacy zip code.
To compare the perception and the spatial accessibility of persons with haemophilia and other coagulation deficiencies regarding prophylactic and on-demand antihemorrhagic treatment | Through study completion, on average 6 months.
  The mean distances between the 4-groups of satisfaction level are compared using an analysis of variance (ANOVA).

SECONDARY OUTCOMES:
To determine if the severity of the disease would be a factor for encouraging or limiting the perception of accessibility to prophylactic or on-demand anti-haemorrhagic treatments | Through study completion, on average 6 months.
  The satisfaction level of participants are stratified on the severity of the disease (minor, moderate, major).
To determine if the age of the patient would be a factor for encouraging or limiting the perception of accessibility to prophylactic or on-demand anti-haemorrhagic treatments | Through study completion, on average 6 months.
  The satisfaction level of participants are stratified on the age of patient.
To determine if the condition of access to hospital would be a factor for encouraging or limiting the perception of accessibility to prophylactic or on-demand anti-haemorrhagic treatments | Through study completion, on average 6 months.
  The satisfaction level of participants are stratified on the condition of access to hospital (relative to traffic conditions, the physical condition of the patient, the parking difficulties).
To determine if the level of autonomy of the participant would be a factor for encouraging or limiting the perception of accessibility to prophylactic or on-demand anti-haemorrhagic treatments | Through study completion, on average 6 months.
  The satisfaction level of participants are stratified on the level of autonomy of the participant (relative to wheelchair, crutch/walking stick or other mobility aid).
To determine if the availability of the hospital pharmacy would be a factor for encouraging or limiting the perception of accessibility to prophylactic or on-demand anti-haemorrhagic treatments | Through study completion, on average 6 months.
  The satisfaction level of participants are stratified on the availability of the hospital pharmacy (relative to the waiting times).

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Fraticelli, PhD, Study Director — RESCUe-RESUVal; Julie Freyssenge, PhD, Study Director — RESCUe-RESUVal
Locations (34):
- France (34):
  - Centre Hospitalier Albertville-Moûtiers, Albertville
  - Centre Hospitalier Annecy Genevois, Annecy
  - Centre Hospitalier d'Ardèche Nord, Annonay
  - Centre Hospitalier d'Ardèche Méridionale, Aubenas
  - Centre Hospitalier Henri Mondor d'Aurillac, Aurillac
  - Centre Hospitalier de Belley, Belley
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - Centre hospitalier de Bourg St Maurice, Bourg-Saint-Maurice
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - Groupement Hospitalier Est, Hospices Civils de Lyon, Bron
  - Centre Hospitalier de Chambéry - Hôpital Savoie, Chambéry
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Hôpital Nord Ouest de Villefranche-sur-Saône, Gleizé
  - Centre Hospitalier Universitaire Grenoble - Alpes, La Tronche
  - Hôpital Edouard herriot, Hospices Civils de Lyon, Lyon
  - Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Centre Hospitalier du Forez, Montbrison
  - Centre Hospitalier de Montélimar, Montélimar
  - Hôpital de Montluçon, Montluçon
  - Centre Hospitalier de Moulins-Yzeure, Moulins
  - Centre Hospitalier Du Haut Bugey, Oyonnax
  - Centre Hospitalier des Vals d'Ardeche, Privas
  - Centre Hospitalier de Roanne, Roanne
  - Hôpitaux Drôme Nord, Romans-sur-Isère
  - Pharmacie Centrale, Hospices Civils de Lyon, Saint-Genis-Laval
  - Centre Hospitalier Intercommunal Sud-Léman Valserine, Saint-Julien-en-Genevois
  - Centre Hospitalier Uuniversitaire Nord, Saint-Étienne, Saint-Priest-en-Jarez
  - Hôpitaux du Pays du Mont-Blanc, Sallanches
  - Hôpital Nord-Ouest Tarare-Grandris, Tarare
  - Hopitaux du Léman, Thonon-les-Bains
  - Centre Hospitalier de Valence, Valence
  - Centre Hospitalier de Vichy, Vichy
  - Centre Hospitalier Lucien Hussel, Vienne

IPD SHARING:
Plan to Share IPD: No
Patient information is held under legal and ethical obligations of confidentiality. As the disease is rare, information should not be used or disclosed in a form that might identify a patient without his or her consent.

REFERENCES:
- [Background] Leroy V, Freyssenge J, Renard F, Tazarourte K, Negrier C, Chamouard V. Access to treatment among persons with hemophilia: A spatial analysis assessment in the Rhone-Alpes region, France. J Am Pharm Assoc (2003). 2019 Nov-Dec;59(6):797-803. doi: 10.1016/j.japh.2019.07.006. Epub 2019 Aug 9. PMID 31405805
- [Background] Susen S, Gruel Y, Godier A, Harroche A, Chambost H, Lasne D, Rauch A, Roullet S, Fontana P, Goudemand J, de Maistre E, Chamouard V, Wibaut B, Albaladejo P, Negrier C. Management of bleeding and invasive procedures in haemophilia A patients with inhibitor treated with emicizumab (Hemlibra(R) ): Proposals from the French network on inherited bleeding disorders (MHEMO), the French Reference Centre on Haemophilia, in collaboration with the French Working Group on Perioperative Haemostasis (GIHP). Haemophilia. 2019 Sep;25(5):731-737. doi: 10.1111/hae.13817. Epub 2019 Jul 11. PMID 31294904